CLINICAL TRIAL: NCT01466985
Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiretroviral Activity of MK-1439 in HIV-1 Infected Patients
Brief Title: A Study of Doravirine (MK-1439) in Human Immunodeficiency Virus Type 1 (HIV-1)-Infected Participants (MK-1439-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1439-005; 2011-003508-19 (EudraCT Number); MK-1439-005 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — doravirine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel A: Doravirine 25 mg or Placebo (Experimental): Participants will receive oral doses of doravirine 25 mg or placebo once daily for 7 days.
  Interventions: Drug: Doravirine; Drug: Placebo
- Panel B: Doravirine 200 mg or Placebo (Experimental): Panel B (doravirine 200 mg or placebo once daily for 7 days) will initiate upon satisfactory review of safety and tolerability from Panel A, and all safety, tolerability and pharmacokinetic data from the study MK-1439-001.
  Interventions: Drug: Doravirine; Drug: Placebo
- Panel C: Doravirine or Placebo (Experimental): Panel C is optional. If conducted, the dose will be confirmed after review of data from prior panels.
  Interventions: Drug: Doravirine; Drug: Placebo

INTERVENTIONS:
Drug: Doravirine — Doravirine tablets, orally, once daily for 7 days at a dose of 25 mg in Panel A and 200 mg in Panel B; dose in Panel C to be determined (≤200 mg).
  Other Names: MK-1439
Drug: Placebo — Placebo tablets once daily for 7 days.

SUMMARY:
This is a study to evaluate the safety, tolerability, pharmacokinetics, and antiretroviral activity of doravirine (MK-1439) as monotherapy in antiretroviral therapy (ART)-naïve, HIV-1-infected participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV-1-infection ≥3 months prior to screening
* Participants with female partner(s) of child-bearing potential must agree to use a medically acceptable method of contraception during the study and for 90 days after the last dose of study drug
* Body Mass Index (BMI) ≤35 kg/m^2
* Other than HIV infection, participant's baseline health is judged to be stable
* No clinically significant abnormality on electrocardiogram (ECG)
* Participant is ART-naïve (defined as having never received any antiretroviral agent or ≤30 consecutive days of an investigational antiretroviral agent (excluding an Non-Nucleoside Reverse Transcriptase Inhibitor [NNRTI]) or ≤60 consecutive days of combination ART not including an NNRTI)
* Participant is willing to receive no other ART for the duration of the treatment phase of this study.

Exclusion Criteria:

* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological (outside of HIV-1 infection), renal, respiratory, or genitourinary abnormalities or diseases
* History of clinically significant neoplastic disease
* Participant has used any immune therapy agents or immunosuppressive therapy within 1 month prior to treatment in this study
* Participant has one or more pre-existing risk factors for Torsades de Pointes (New York Heart Association Functional Classification II through IV heart failure, familial long-QT-syndrome, uncorrected hypokalemia, QTcF >470 msec)
* Participant requires or is anticipated to require chronic daily prescription medications
* Current (active) diagnosis of acute hepatitis due to any cause
* History of chronic Hepatitis C virus (HCV) unless there has been documented cure and/or patient with a positive serologic test for HCV has a negative HCV viral load.
* Positive Hepatitis B surface antigen
* Participant is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort [Hypericum perforatum]) beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study, until the post-study visit
* Participant consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Participant consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Participant is an excessive smoker (i.e., more than 10 cigarettes/day) and is unwilling to restrict smoking to ≤10 cigarettes per day
* Major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit
* Participation in another investigational study within 4 weeks prior to the prestudy (screening) visit
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Current regular user (including use of any illicit drugs) or has a history of drug (including alcohol) abuse within approximately 1 year

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10-21 (Actual); Primary Completion 2012-04-10 (Actual); Study Completion 2012-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Schurmann D, Sobotha C, Gilmartin J, Robberechts M, De Lepeleire I, Yee KL, Guo Y, Liu R, Wagner F, Wagner JA, Butterton JR, Anderson MS. A randomized, double-blind, placebo-controlled, short-term monotherapy study of doravirine in treatment-naive HIV-infected individuals. AIDS. 2016 Jan 2;30(1):57-63. doi: 10.1097/QAD.0000000000000876. PMID 26372481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with human immunodeficiency virus type 1 (HIV-1) who were antiretroviral therapy (ART)-naïve were enrolled at a single study center in Germany.
Pre-assignment Details: Participants were allocated into panels, then randomized to doravirine 25 mg or placebo (Panel A) or doravirine 200 mg or placebo (Panel B). The protocol planned for a possible Panel C but Panel C was not enrolled. Study results are presented according to actual treatment received.
Groups:
- Doravirine 25 mg: Participants with HIV-1 infection received doravirine 25 mg q.d. for 7 days.
- Doravirine 200 mg: Participants with HIV-1 infection received doravirine 200 mg q.d. for 7 days.
- Placebo: Participants with HIV-1 infection received placebo q.d. by mouth for 7 days.
Period: Overall Study
Arm/Group | Doravirine 25 mg | Doravirine 200 mg | Placebo
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doravirine 25 mg | Doravirine 200 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (5.8) | 34.8 (8.4) | 26.8 (1.0) | 32.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in HIV-1 Ribonucleic Acid (RNA) Viral Load
Description: The change from baseline to Day 7 in plasma HIV RNA viral load was determined for each arm. Results are expressed as change in HIV RNA log10 copies/mL after 7 daily doses of doravirine or placebo. It was hypothesized that at least 1 dose of doravirine would be superior to placebo as documented by the upper bound of the 90% confidence interval <-1. Plasma HIV RNA levels were determined using the Abbott RealTime HIV assay which has a linear range from 40 to 10 million copies/mL.
Time Frame: Baseline and Day 7
Population: All participants who received ≥1 dose of study drug are included (results are presented according to actual treatment received).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Doravirine 25 mg | Doravirine 200 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6
Percentage change | -1.52 [-1.71 to -1.32] | -1.41 [-1.61 to -1.21] | -0.15 [-0.35 to 0.06]
Statistical Analysis 1: Comparison: Doravirine 25 mg vs Placebo; Test type: Superiority — Doravirine was declared superior to placebo when the upper bound of the 90% CI was <-1; p < 0.001, ANCOVA; Least squares (LS) mean difference = -1.37, 90% CI [-1.60 to -1.02]
Statistical Analysis 2: Comparison: Doravirine 200 mg vs Placebo; Test type: Superiority — Doravirine was declared superior to placebo when the upper bound of the 90% CI was <-1; p < 0.001, ANCOVA; LS mean difference = -1.26, 90% CI 2-sided [-1.51 to -1.02]

2. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Dosing to 24 Hours Postdose (AUC0-24hr) of Doravirine on Day 7
Description: The AUC0-24hr of doravirine on Day 7 was determined in the doravirine treatment arms.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12 and 24 hours postdose on Day 7
Population: All participants who received ≥1 dose of doravirine are included.
Measure: Geometric Mean (90% Confidence Interval); unit: uM*hr
Arm/Group | Doravirine 25 mg | Doravirine 200 mg
Number analyzed (Participants) | 6 | 6
uM*hr | 11.2 [9.35 to 13.4] | 62.2 [52.0 to 74.4]

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Doravirine on Day 7
Description: The Cmax of doravirine on Day 7 was determined in the doravirine treatment arms.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12 and 24 hours postdose on Day 7
Population: All participants who received ≥1 dose of doravirine are included.
Measure: Geometric Mean (90% Confidence Interval); unit: nM
Arm/Group | Doravirine 25 mg | Doravirine 200 mg
Number analyzed (Participants) | 6 | 6
nM | 826 [727 to 938] | 4300 [3790 to 4890]

4. Secondary Outcome: Plasma Concentration 24 Hours Postdose (C24hr) of Doravirine on Day 7
Description: The C24hr of doravirine on Day 7 was determined in the doravirine treatment arms.
Time Frame: 24 hours postdose on Day 7 (Day 8)
Population: All participants who received ≥1 dose of doravirine are included.
Measure: Geometric Mean (90% Confidence Interval); unit: nM
Arm/Group | Doravirine 25 mg | Doravirine 200 mg
Number analyzed (Participants) | 6 | 6
nM | 251 [188 to 335] | 1540 [1150 to 2060]

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Doravirine on Day 7
Description: The Tmax of doravirine on Day 7 was determined in the doravirine treatment arms.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12 and 24 hours postdose on Day 7
Population: All participants who received ≥1 dose of doravirine are included.
Measure: Median (Full Range); unit: Hours
Arm/Group | Doravirine 25 mg | Doravirine 200 mg
Number analyzed (Participants) | 6 | 6
Hours | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 4.00]

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug (up to 21 days)
Description: All participants who received ≥1 dose of study therapy are included. Adverse event d are summarized by study treatment received for the 7-day treatment period and are pooled for the 14-day poststudy period.
Groups:
- Poststudy: AEs from all participants in the study were pooled for the poststudy period.
Arm/Group | Doravirine 25 mg | Doravirine 200 mg | Placebo | Poststudy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/18
Other Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 3/6 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine 25 mg (N=6) | Doravirine 200 mg (N=6) | Placebo (N=6) | Poststudy (N=18)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine 25 mg (N=6) | Doravirine 200 mg (N=6) | Placebo (N=6) | Poststudy (N=18)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsilitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.